CLINICAL TRIAL: NCT03052114
Title: Imaging Stroke, Epilepsy and Evoked Potentials in the Brain Using Electrical Impedance Tomography
Brief Title: Electrical Impedance Tomography of Stroke and Brain Injury
Status: Active, not recruiting | Type: Observational
Sponsor: University College, London (Other)
Collaborators: University College London Hospitals (Other)
Responsible Party: Sponsor
Other Study IDs: 14/0861b
Record Dates: First submitted 2017-02-09; First posted 2017-02-14 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Stroke; Craniocerebral Injuries
Keywords: Electrical Impedance Tomography; EIT; Stroke; Craniocerebral Injury; Head Injury
MeSH Terms: conditions — Stroke; Craniocerebral Trauma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Stroke: Electrical Impedance Tomography with scalp electrodes
  Interventions: Device: Electrical Impedance Tomography
- Head Injury: Electrical Impedance Tomography with scalp electrodes
  Interventions: Device: Electrical Impedance Tomography

INTERVENTIONS:
Device: Electrical Impedance Tomography — EIT comprises of a box of electronics similar in size to a video recorder, laptop computer and leads which link typically to 16 or 32 external ECG-like electrodes placed around the subject. Images are generated by applying tiny electrical signals through some electrodes and recording the resulting signals at others. The signals applied are completely safe, within established British and EU safety limits and cannot be felt.
  Other Names: EIT

SUMMARY:
The purpose of this study is to determine if Electrical Impedance Tomography (EIT) can produce reproducible and accurate images in people with stroke or head injury compared to existing standards such as MRI, CT.

Electrical Impedance Tomography is a relatively new medical imaging method, which has the potential to provide novel images of brain function. It is fast, portable, safe and inexpensive, but currently has a relatively poor spatial resolution. It produces images of the internal electrical impedance of a subject with stroke or head injury using rings of ECG like electrodes on the skin. EIT recording will take place as early as possible, usually within 24 hours of admission. Following completion of the recording, the EIT images will subsequently be analysed and compared to other imaging data for accuracy.

DETAILED DESCRIPTION:
Electrical Impedance Tomography (EIT) is a novel medical imaging method in which tomographic images are rapidly produced using electrodes placed around the body. The principal applicant's group has demonstrated that EIT can rapidly image functional brain activity in stroke, epilepsy and normal activity in animal models and has developed instrumentation and image reconstruction algorithms which work well in head-shaped tanks.

The principal aim of this research is to optimise and assess accuracy of Electrical Impedance Tomography (EIT) using scalp electrodes in imaging stroke/head injury in human participants. EIT could provide a unique new imaging modality which could provide continuous monitoring at the bedside after head injury or diagnosis in the back of an ambulance or GP surgery and so permit rapid deployment of thrombolytic therapy. If successful, EIT would become a standard imaging technique available in all ambulances and A&E departments for this purpose. It would be used in all cases of suspected stroke which present except to dedicated acute stroke centres. Imaging could be undertaken at presentation by paramedical staff if in an ambulance, or nurses or radiographers if in A&E. Images would be reported by radiologists remotely who could then sanction administration of thrombolytic agents by physicians, nurses or paramedical staff. EIT would allow neuroimaging to be undertaken significantly earlier in all situations where a dedicated stroke centre with available urgent CT was not available. This would benefit clinical staff who could provide an improved service and patients, who would enjoy improved outcome and greater access to thrombolytic therapy.

The recording will take place with scalp electrodes while the patient sits comfortably in a chair or lies on a bed. Recording takes for 10 minutes to 1 hour. In some subjects, EIT can be used to image changes in the brain over hours following head injury. In this case, recording will take place over hours or days with scalp electrodes according to the clinical situation. Stroke patients could also be recorded in this study, as similar changes in the injured brain could also occur after stroke. Following completion of the recording, scalp electrodes and any paste will be removed. Collected data will be analysed and compared to other imaging data.

ELIGIBILITY:
Inclusion Criteria:

* Patient with MRI or CT evidence of a stroke
* Ability to give informed consent or have a consultee able to provide informed consent (for stroke group)
* Any subject admitted for observation following a head injury (for head injury group)

Exclusion Criteria:

* non (for stroke group)
* Any skull fractures or other injury which precludes the safe application of scalp electrodes (for head injury group)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke patients or patients under hospital observation after a head injury at the University College Hospital
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2015-10; Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
EIT images accuracy | three years
  images accuracy defined by the image errors

CONTACTS AND LOCATIONS:
Overall Officials: David S Holder, Professor, Principal Investigator — University College London, University College Hospital
Locations (1):
- Hyper-Acute Stroke Unit University College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided